CLINICAL TRIAL: NCT06811064
Title: Resource Parents in Neonatology: Innovative Partnership Practices to Improve Quality of Life After Returning Home
Brief Title: Involving Family Stakeholders in the NICU: a New Perspective to Improve Quality of Life. PAREN
Acronym: PAREN
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A01087-36
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Premature Birth
Keywords: resource parents; quality of life; premature newborn; neonatal intensive care unit
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Intervention of resource parents for parents of hospitalised premature new born: Parents of hospitalised premature new born watch a testimony video pf other parent who experienced hospitalization of their premature new born
  Interventions: Other: Testimony video
- without intervention of resource parents for parents of hospitalised premature new born: Parents of hospitalised premature new born do not watch a testimony video of other parent who experienced hospitalization of their premature new born

INTERVENTIONS:
Other: Testimony video — A testimonial video on the experiences of parents of premature babies during the transfer of their newborn from the intensive care unit to the neonatal unit. This video will be performed with the collaboration of the carers and resource parents.
  Groups: Intervention of resource parents for parents of hospitalised premature new born

SUMMARY:
Introduction Thanks to medical advances in neonatal care, the majority of children admitted to the neonatal intensive care unit (NICU) survive and enjoy a good quality of life. At the same time, medical practices and philosophy of neonatal care have changed and families are playing an increasingly important role in their child's care. However, stress and anxiety generated by hospitalization and complex technologies of neonatal intensive care units may be an obstacle to integrate parents and help them take ownership of their role. A number of measures have been established to improve the experience of parents in neonatology, such as multidisciplinary care, involving psychologists, social workers, spiritual care workers, psychomotor therapists and physiotherapists.

Among these interventions, the introduction of resource parents (RPs), parents who have previously been involved in neonatology, is a new initiative that is growing rapidly in North America. These RPs bring a unique perspective based on their experiential knowledge. This partnership model is still underdeveloped in France, and its impact on parents' quality of life and early interactions with their children has been little studied or described.

Method Our aim is therefore to develop a PR intervention in neonatology units and measure its impact in the short and medium term, with a prospective multicenter step wedge study.

The chosen intervention will be co-constructed with PRs. It will take the form of testimonial videos focusing on one of the key moments in the care of newborn babies: the transition from different neonatology units. These videos will then be viewed by parents of hospitalized newborn in the units at the time of their transition. A survey assessing the parents' Self Perceived Efficacity in taking care of their child will be administered when the child transitions to the neonatal unit and then again when the child is discharged from the hospital. At the one-year old visit, the families' quality of life will be assessed using another standardized survey: the Pediatric Quality of Life Inventory (PedsQLTM2.0) - Family Impact Module.

Perspective Our hypothesis is that a PR intervention at a key point in the newborn's care pathway can help parenthood and have a positive impact on early interactions and quality of life at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Premature newborn (<37 weeks of amenorrhoea)
* Newborn whose parents are aged 18 or over
* Newborns who have spent at least one week in a neonatal intensive care unit,
* Newborn baby hospitalised in one of the neonatology/intensive care unit
* Newborn for whom both or one of the two parents have expressed their non-opposition to taking part in the study or Newborn for whom the only legal representative (single-parent family) has expressed his/her non-opposition to taking part in the study.

Exclusion Criteria:

* Newborns at term (≥ 37 SA);
* Newborns in which both or one of the parents refuse to participate or newborns in which the only legal representative (single-parent family) has expressed opposition to participating in the study.
* Newborn whose two parents or one of them withdraws their non-opposition
* Newborn transferred to another neonatal intensive care unit during hospital stay;
* Newborn child who dies during hospitalisation or after discharge up to the one-year visit.
* Newborn lost to follow-up at 1 year.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: premature newborn
Sampling Method: Non-Probability Sample
Enrollment: 1008 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Evaluate the the quality of life of parent with premature child at one year corrected age | At the one year anniversary (12 months corrected age) of the premature child
  Questionnaire PedsQL

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde LEFEVRE, Study Director — assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique des Hôpitaux de Marseille (APHM), Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided